CLINICAL TRIAL: NCT06821360
Title: Evaluating the Practicalities & Potential Benefits of Using Remote C-peptide Testing in Clinical Practice to Confirm Established Type 1 Diabetes
Brief Title: Assessing Remote Confirmation of Type 1 Diabetes
Acronym: ARC-T1D
Status: Enrolling by invitation | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: NIHR Exeter Clinical Research Facility (Network); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: 338864; 2410662 (Other: Royal Devon University Healthcare NHS Foundation Trust)
Record Dates: First submitted 2025-02-10; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Type 1 Diabetes (T1D)
Keywords: Diabetes diagnosis. Insulin levels. Remote testing. C-peptide. Home finger-prick samples.
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Cohort: Adults treated as Type 1 diabetes (T1D) and under the clinical care of the specialist diabetes team(s) at the Royal Devon University Healthcare NHS Foundation Trust. Diabetes duration >3 years at the time of study participation. Aged > 18 at the time of study participation.
  Interventions: Diagnostic Test: C-peptide test

INTERVENTIONS:
Diagnostic Test: C-peptide test — Participants collect a single home finger-prick sample and post to the clinical laboratory for C-peptide analysis (a measure of endogenous insulin production).

SUMMARY:
The aim of this research is to assess the practicalities and potential benefits of collecting home finger prick samples from all patients within a hospital type 1 diabetes service to test how much insulin each patient is producing. To do this we will send detailed study information, sample collection kits and reply-paid return packs to 1500 randomly selected patients, treated as type 1 diabetes, in a hospital clinic (3000 patients in the whole clinic). We will ask participants to consent to take part (either online or by completing a paper consent form returned with their pack) before collecting a finger prick blood sample. We will ask participants to collect the sample between 1 and 5 hours after a meal and to check and record their blood glucose level at the same time. Participants will then return the sample and glucose result, using the pre-paid pack provided, to the hospital clinic laboratory for a test called C-peptide (a measure of how much of their own insulin they are producing). The sample collection process should take no longer than 10 minutes.

We will record the percentage of patients returning samples within 4 weeks of initial contact and determine the number of cases with high C-peptide suggestive of non-type 1 diabetes. If this study shows remote C-peptide testing is a practical and acceptable to patients, it could allow this remote service to be offered to all type 1 diabetes clinics in every hospital in the United Kingdom. An estimated 350,000 people in the United Kingdom have type 1 diabetes. Reclassifying an estimated 1 in 15 people would mean approximately 23,000 people nationally could benefit from being identified as potentially able to stop insulin treatment.

DETAILED DESCRIPTION:
Background It can be hard to diagnose type 1 diabetes in adults because the symptoms can overlap with type 2 diabetes and misclassification of type 2 and type 1 diabetes can occur. This matters as type 2 diabetes cases misclassified as having type 1 diabetes potentially receive a lifetime of unnecessary insulin treatment without access to the effective treatment strategies for type 2 diabetes. Whether someone needs treating as type 1 diabetes can be confirmed by measuring their insulin levels using a test called C-peptide. This should be measured when diabetes is longstanding (over 3 years diabetes duration) as, at diagnosis levels of insulin secretion can overlap in type 1 and type 2 diabetes. A study in Scotland measured C-peptide in a clinic of patients with long standing treatment as type 1 diabetes showing around 1 in 15 of cases did not have type 1 diabetes.

As a result, in Scotland all those with longstanding type 1 diabetes now have C-peptide measured and this is likely to be recommended across the UK. For newly diagnosed cases this will occur prospectively as part of patients' ongoing type 1 diabetes care. However, for existing cases, each hospital will need to test C-peptide, on a blood sample collected from a vein, in all patients in their type 1 diabetes clinic. In addition to the burden on clinical staff to collect the samples, this C-peptide test is not measured in many UK laboratories so co-ordinating this testing on all patients within a clinic will be extremely challenging.

We have recently validated a method of testing C-peptide on capillary blood (finger prick) samples. Importantly these can be collected by a patient at their home and can be posted back to any UK laboratory where C-peptide measurement is available. Using this approach means that clinic visits for blood collection are not required and testing can be co-ordinated from a central location, making organising testing in a whole clinic much more straightforward.

Study Aims & Participation The aim of this research is to assess the practicalities & potential benefits of collecting home finger prick samples from all patients within a hospital type 1 diabetes service to test how much insulin each patient is producing. To do this we will send detailed study information, sample collection kits and reply-paid return packs to 1500 randomly selected patients from a type 1 diabetes clinic (3000 patients in the whole clinic). We will ask participants to consent to take part (either online or by completing a paper consent form returned with their pack) before collecting a finger prick blood sample. We will ask participants to collect the sample between 1 and 5 hours after a meal and to check and record their blood glucose level at the same time. Participants would then return the sample and glucose result, using the pre-paid pack provided to the hospital clinic laboratory for a test called C-peptide (a measure of how much of their own insulin a person is producing). The sample collection process should take no longer than 10 minutes.

We will record the percentage of patients returning samples within 4 weeks of initial contact and determine the number of cases with high C-peptide suggestive of non-type 1 diabetes. If this study shows remote C-peptide testing is practical, and acceptable to patients, it could lead to remote testing being offered at all type 1 diabetes clinics in every hospital in the United Kingdom. Diabetes UK estimates around 350,000 people in the United Kingdom have type 1 diabetes. Reclassifying 1 in 15 people would mean approximately 23,000 people nationally could benefit from being identified as potentially able to stop insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Type 1 diabetes follow up code OR rapid progression to insulin (within 3 years of diagnosis) to capture miscoded cases.
* Under the clinical care of the diabetes team(s) at the Royal Devon University Healthcare NHS Foundation Trust
* Duration of diabetes >3 years
* Aged 18 years or older.

Exclusion Criteria:

* Patients considered by their clinical care team to be unsuitable/inappropriate to be invited to take part in this research (e.g. severe sight impairment, reduced capacity to consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Type 1 diabetes follow up code OR rapid progression to insulin (within 3 years of diagnosis) to capture miscoded cases. Under the clinical care of the diabetes team(s) at the Royal Devon University Healthcare NHS Foundation Trust
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-03 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of samples returned | Within 4 weeks of initial contact
  The number of completed samples returned within four weeks of sample pack mailout.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Thomas, PhD MRCP, Principal Investigator — University of Exeter and Royal Devon University Healthcare NHS Foundation Trust
Locations (1):
- NIHR Exeter Clinical Research Facility, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No